CLINICAL TRIAL: NCT05970198
Title: A Prospective Randomized Controlled Study of Helical Tomotherapy for Pre-transplantation Pretreatment of Autologous Hematopoietic Stem Cells in Multiple Myeloma
Brief Title: Helical Tomotherapy in Multiple Myeloma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fuling Zhou (Other)
Responsible Party: Sponsor-Investigator, Fuling Zhou, Chief physician, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08
Record Dates: First submitted 2023-07-12; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autologous hematopoietic stem cell transplantation (Active Comparator): Porting method melphalan: recommended dose of 70 mg/m2/day with 2 consecutive days (days -2 and -1) intravenous (IV) for more than 30 minutes each prior to autologous hematopoietic stem cell transplantation (ASCT, day 0).
  Interventions: Procedure: Autologous hematopoietic stem cell transplantation
- Radiotherapy combined with autologous hematopoietic stem cell transplantation (Experimental): TMI radiation dose On the 5th day (-5 days) before transplantation, an irradiation dose of 8 Gy is given.
  TMI uses a 6-18MV linear accelerator, the patient lies on his side in a single irradiation field, covered with a 1 cm thick plexiglass frame, and the radioactive source is 4 meters away from the body surface of the human side. The anterior and anterior positions were alternately irradiated, and the horizontal beam was irradiated in the opposite direction, and the actual irradiation dose was detected by the thermo-optical element of the 2570 roentgen dosimeter scale, and the irradiation dose of all parts of the body was adjusted to make the abdominal irradiation dose difference within 10%, the total dose was 8Gy, divided into 2 times a day, with an interval of 5 hours, and the dose rate was 4.99-6.96cGy/min.Porting method melphalan.
  Interventions: Radiation: Total Marrow irradiation，TMI; Procedure: Autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Radiation: Total Marrow irradiation，TMI — TMI radiation dose On the 5th day (-5 days) before transplantation, an irradiation dose of 8 Gy is given.
  TMI uses a 6-18MV linear accelerator, the patient lies on his side in a single irradiation field, covered with a 1 cm thick plexiglass frame, and the radioactive source is 4 meters away from the body surface of the human side. The anterior and anterior positions were alternately irradiated, and the horizontal beam was irradiated in the opposite direction, and the actual irradiation dose was detected by the thermo-optical element of the 2570 roentgen dosimeter scale, and the irradiation dose of all parts of the body was adjusted to make the abdominal irradiation dose difference within 10%, the total dose was 8Gy, divided into 2 times a day, with an interval of 5 hours, and the dose rate was 4.99-6.96cGy/min.
  Arms: Radiotherapy combined with autologous hematopoietic stem cell transplantation
Procedure: Autologous hematopoietic stem cell transplantation — Autologous hematopoietic stem cell transplantation;Porting method melphalan

SUMMARY:
To explore the safety and efficacy of systemic radiotherapy (TBI) combined with melphalan (Mel) for pretreatment of autologous hematopoietic stem cells in multiple myeloma.

DETAILED DESCRIPTION:
This study is a single-center, prospective clinical study targeting myeloma patients requiring transplantation, and investigating the efficacy and safety of TBI combined with Mel regimen for transplant pretreatment. Subjects who meet the enrollment criteria were screened to enter the study and receive the corresponding regimen treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Multiple myeloma patients receiving induction therapy and stem cell mobilization preparation for autologous transplantation;
2. Should agree to comply with all contraceptive requirements; 3, ECOG≤2;

4. Total bilirubin, ALT and AST <2×UNL (upper limit of normal), BUN < 30 mg/dL; 5. At least 2 x 10^6 CD34+ cells /kg were collected; 6.absolute neutrophil count >1000/uL and a platelet count of >100,000/uL; 7. The expected survival time is more than 3 months; 8. Written informed consent was obtained from the patients or their immediate family members.

Exclusion Criteria:

Any of the following was an exclusion criterion:

1. According to the investigator's judgment, patients who cannot tolerate melphalan and radiotherapy;
2. Patients with known active hepatitis B virus (HBV) or hepatitis C virus (HCV), or seropositive for human immunodeficiency virus (HIV);
3. patients with uncontrolled or severe cardiovascular disease
4. According to the protocol or the investigator's judgment, the patient has a serious physical or mental illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate and above 100 days after transplantation (≥ CR rate) | through study completion, an average of 1 year
  Complete response rate and above 100 days after transplantation (≥ CR rate)

SECONDARY OUTCOMES:
1-year Progression-free Survival rate | 1 year
  1-year Progression-free Survival rate

OTHER OUTCOMES:
1-year Overall Survival rate | 1 year
  1-year Overall Survival rate
Platelet implantation time | 3 months
  Platelet implantation time
Neutrophil implantation time | 3 months
  Neutrophil implantation time

CONTACTS AND LOCATIONS:
Overall Officials: Fuling Zhou, Study Director — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No